CLINICAL TRIAL: NCT06789588
Title: Pharmacogenetic Algorithm for Warfarin Dose Predictor: Protocol for Improvement and Effectiveness of Therapy Anticoagulant
Brief Title: Protocol for Improvement of Therapy With Warfarin
Acronym: WARFALGORIT
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pernambuco (Other)
Collaborators: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Maria Mariana Barros Melo Da Silveira, PhD, University of Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 77321024.4.0000.5192; 444198/2023-7 (Other Grant/Funding Number: Conselho Nacional de Desenvolvimento Científico e Tecnológico)
Record Dates: First submitted 2025-01-17; First posted 2025-01-23 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF)
Keywords: atrial fibrillation; oral anticoagulant; warfarin; genetic polymorphism
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Group 1 (Intervention): Patients with AF using or indicating the need to start OAC therapy guided by a pharmacogenetic algorithm that predicts the dose of warfarin.
  Group 2 (control): Patients with AF indicated for OAC therapy guided by institutional protocol.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 Experimental (Experimental): Patients with AF using or indicating the need to start OAC therapy guided by a pharmacogene
  Interventions: Drug: pharmacogenetic algorithm
- Group 2 Active Comparator (Active Comparator): Patients with AF indicated for OAC therapy guided by institutional protocol.
  Interventions: Drug: Clinical treatment

INTERVENTIONS:
Drug: pharmacogenetic algorithm — The dose predictor algorithm proposed in this work aims to maintain and quality treatment in an individualized and effective manner. In the routine use protocol, warfarin is prescribed based only on the INR collected within 5 days. The proposed intervention protocol is based on the patient's clinical and genetic factors, such as genetic polymorphisms, age, weight, height, race, use of amiodarone, statins, antifungals or antibiotics, tobacco use, clinical indication and what the RNI target.
  Arms: Group 1 Experimental
Drug: Clinical treatment — Patients with AF indicated for OAC therapy guided by institutional protocol.
  Arms: Group 2 Active Comparator

SUMMARY:
Atrial Fibrillation (AF) is the most common supraventricular arrhythmia in clinical practice. The presence of AF, as an independent factor, increases mortality by up to two times. One in every six cerebrovascular accidents (CVA) occurs in patients with AF, generating an annual risk of around 7% per year, which represents an increase of up to seven times in relation to the risk in the general population, leading to the need for start anticoagulant therapy. Warfarin is still the Oral Anticoagulant (OC) of choice, being the most used in several clinical situations. The variability of response to anticoagulants is related to pharmacokinetic and pharmacodynamic factors, adherence to treatment, age, diet, body mass index (BMI), liver function, body deposition of vitamin K, individual drug metabolism, drug interactions, comorbidities, in addition to of genetic factors. It is estimated that the annual risks associated with the use of OCs are between 2% and 8% for bleeding. The clinical benefit and risk of OAC therapy are associated with the time in which the values of therapeutic - TTR (time in therapeutic range). Measuring the quality of anticoagulation assesses whether therapy is being maintained within this range. Increased TTR is associated with a decrease in thromboembolic and/or hemorrhagic events. In the context of OCs, pharmacogenetics is the science that predicts the response to drugs, based on individual genetic markers. By understanding the relationship between the genotype and the response to a drug, pharmacogenomics has the potential to help healthcare professionals to predict the therapeutic dose of warfarin by genotyping patients for several Single Nucleotide Polymorphisms (SNPs) that affect metabolism or sensitivity to warfarin. Therefore, the main objectives of genotype-guided therapy are to improve the safety and efficacy of anticoagulant therapy. In Brazil, more specifically in the Brazilian Northeast, the use of a dose predictor algorithm is not common, which leads to high rates of complications and consequently increases the length of hospital stay. As a result, there is an increasing need to implement therapeutic technologies applied to precision health, explore studies on genetic polymorphisms and therapies guided by pharmacogenomics, aiming to understand the individual genetic effect on the metabolism of drugs such as warfarin.

DETAILED DESCRIPTION:
Atrial Fibrillation (AF) is the most common supraventricular arrhythmia in clinical practice. Patients with AF have a 5 times greater risk of causing stroke, especially ischemic stroke, than any other cardiovascular disease. This arrhythmia causes stasis and changes in the thrombosis-antithrombosis balance, which can form thrombi and embolize systemically, reaching the brain and causing stroke, leading to the need to start anticoagulant therapy. Warfarin is still the Oral Anticoagulant (OAC) of choice, being the most used in various clinical situations. With sensitivity to the drug varying in each person, treatment needs to be monitored regularly using the International Normalized Ratio (INR). The known genetic variants that have the greatest impact on the response to warfarin are the variants in the warfarin target, VKORC1, carriers of this variant require a lower dose of warfarin, and the enzyme encoded by CYP2C9, which is the most important when it comes to of involvement with the pharmacokinetics of warfarin. Polymorphisms in the CYP2C9 and VKORC1 genes are responsible for approximately 12 and 24%, respectively, of the variation in warfarin dose among. patients of European descent. Therefore, in the presence of one or more polymorphisms in one of these genes, it is necessary to adjust the warfarin doses. Previous studies have indicated that pharmacogenetic algorithms generally predict warfarin dose more accurately than other dosing methods. In Brazil, more specifically in the Brazilian Northeast, the use of a dose predictor algorithm is not common, which leads to high rates of complications and consequently increases the length of hospital stay. As an objective, the present study plans to implement a pharmacogenetic algorithm protocol for predicting warfarin dose, guided by genotype, versus a clinical protocol based only on drug dosage, in the population with atrial fibrillation, and to evaluate the superiority of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be greater than or equal to 18 years old
* Patients using warfarin or indicated to start therapy
* Patients with AF in its various etiologies and in paroxysmal, persistent or permanent clinical presentations, with a diagnosis established through clinical examination confirmed by conventional electrocardiographic recording or by 24-hour ambulatory electrocardiographic recording (Holter)

Exclusion Criteria:

* Patients who are not able to understand the explanations about the exams, as well as clarifications inherent to their participation in the research
* Patients who stop following the instructions provided by researchers or whose questionnaires are incomplete;
* Patients with liver disease or cancer of any etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 6 month
  Assess the incidence of adverse events

SECONDARY OUTCOMES:
incidence of adverse events (thromboembolic and hemorrhagic) | 6 month
  clinical evaluation of the decrease of adverse events
Time in therapeutic range | 6 month
  Assess the INR and its time within the therapeutic range

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pernambuco, Recife, Pernambuco, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Respecting the general data protection law of the country of origin (Law No. 13,709/2018), obliterating the data that would identify the participants, we will grant, if necessary, the disclosure of genetic and clinical results, for research purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: January 1, 2027 - January 1, 2032

REFERENCES:
- See also: Study that formed the basis for the current project. — https://pubmed.ncbi.nlm.nih.gov/31447576/
- See also: complementary study — https://pubmed.ncbi.nlm.nih.gov/28198005/